CLINICAL TRIAL: NCT03202212
Title: Effect of Mixed On-line Hemodiafiltration on Circulating Markers of Inflammation and Vascular Dysfunction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Vincenzo Cantaluppi, Principal investigator - Associate Professor of Nephrology, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0030959 CEI/568
Record Dates: First submitted 2017-06-08; First posted 2017-06-28 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Chronic Kidney Failure; Dialysis Related Complication
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: 30 patients treated with a standard 3-time per week bicarbonate high-flux hemodialysis will be randomized 1:1 to continue the treatment or to be switched to mixed on-line hemodiafiltration for 9 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixed on-line hemodiafiltration (Experimental): Mixed on-line hemodiafiltration (mOL-HDF using FX 1000 CorDiax, Fresenius Medical Care, Bad Homburg, Germany), three sessions per week, four hours per session
  Interventions: Procedure: mixed on-line hemodiafiltration
- High flux bicarbonate dialysis (Active Comparator): Standard high flux bicarbonate dialysis with polysulfone membrane, three sessions per week, four hours per session
  Interventions: Procedure: High flux bicarbonate dialysis

INTERVENTIONS:
Procedure: mixed on-line hemodiafiltration — This is a mixed hemodepurative technique exploiting diffusion and convection through a semi-permeable membrane. Dialysis solution is not only interfacing with blood through the membrane (as in bicarbonate hemodialysis) but it is also mixed with it with a pre- and a post- filter dilution. The same amount of fluid added to the bloodstream is then removed within the filter through an appropriate negative pressure in the dialysis solution compartment and thanks a high permeability membrane. Patients will be treated three sessions per week, four hours per session
  Arms: Mixed on-line hemodiafiltration
Procedure: High flux bicarbonate dialysis — Standard high flux bicarbonate dialysis with polysulfone membrane, three sessions per week, four hours per session
  Arms: High flux bicarbonate dialysis

SUMMARY:
On line haemodiafiltration (OL-HDF) has been shown to improve intra-dialytic hemodynamics and cardiovascular outcomes. Several potential candidates of these beneficial effects have been explored. The aim of this study was to investigate the impact of mixed OL-HDF (mOL-HDF) on different circulating mediators of vascular dysfunction.

DETAILED DESCRIPTION:
This is an open label placebo-controlled randomized clinical trial to assess the effect of mixed OL-HDF (mOL-HDF) on different circulating mediators of vascular dysfunction.

Inclusion criteria: age > 18 yrs, hemodialytic treatment from at least 6 months (3 times for week), blood flow rate (Qb) ≥ 250 ml/min using arterovenous fistula (AVF) or permanent central venous catheter (CVC), blood creatinine clearance <5 ml/min, urine output<500 ml/die.

Exclusion criteria: neoplastic diseases, chronic autoimmune diseases, lack of consent, solid organ or bone marrow transplantation.

Safety Assessment: the use of mOL-HDF has been approved by the European Medicines Agency as routine hemodepurative technique for end stage renal disease patients. Patients were evaluated for adverse reaction at each dialysis section; investigators recorded intra and extra-dialytic adverse events.

Study Treatment, Dosage, and Route of Administration: Enrolled patients have been randomized in 2 groups: 15 patients continued high flux bicarbonate hemodialysis (BHD), whereas 15 patients switched to mixed on-line hemodiafiltration (mOL-HDF using FX 1000 CorDiax, Fresenius Medical Care, Bad Homburg, Germany) for 9 months.

Efficacy Assessments:

Main outcome variable: changes in RNA content of circulating exosome/microvesicles (at 9 months) Secondary outcomes: changes in circulating inflammatory markers (C-Reactive Protein, Neutrophil Gelatinase Associated Lipocalin, Interleukin-6, Ferritin) at 3-6 and 9 months. changes in RNA content of circulating microvesicles (at 3 and 6 months)

Study Duration: 9 months

Statistical Methods: Data have been analyzed according to an intention-to-treat approach. Statistical analysis was performed using the unpaired Student t -test, ANOVA, or Kruskal-Wallis test when appropriate. A two-sided value of p=0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* hemodialytic treatment from at least 6 months (3 times for week), blood flow rate during dialysis session (Qb) ≥250 ml/min using arterovenous fistula (AVF) or permanent central venous catheter (CVC), blood creatinine clearance <5 ml/min, urine output <500 ml/die.

Exclusion Criteria:

* neoplastic diseases, autoimmune diseases, solid organ or bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2014-02-10 (Actual); Study Completion 2014-11-11 (Actual)

PRIMARY OUTCOMES:
RNA content of circulating particles | Study start (time 0) and study end (9 months)
  Quantitative micro-RNA changes in plasmatic exosomes/microvesicles assessed by quantitative real-time PCR

SECONDARY OUTCOMES:
Circulating inflammatory markers | All the study timepoints: time 0 and 3, 6, 9 months
  Quantitative changes in C-Reactive Protein, Neutrophil Gelatinase Associated Lipocalin, Interleukin-6, Ferritin
RNA content of circulating particles | All the study timepoints: time 0 and 3, 6, 9 months
  Quantitative micro-RNA changes in plasmatic exosomes/microvesicles assessed by quantitative real-time PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Città della Salute e Della Scienza di Torino - Presidi CTO e Molinette, Torino, To, Italy

IPD SHARING:
Plan to Share IPD: Yes
At the time of registration the study was already completed. IPD data will be available upon request till the study publication, then data will be enclosed within the publication as supplementary material.